CLINICAL TRIAL: NCT04462627
Title: Reduction of COVID 19 Transmission to Health Care Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanane EL KENZ (Other)
Responsible Party: Sponsor-Investigator, Hanane EL KENZ, Head Physician of the Blood Bank, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-BDS-COVID19
Record Dates: First submitted 2020-07-07; First posted 2020-07-08 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Covid 19 positive patients (Experimental)
  Interventions: Diagnostic Test: Blood group determination; Diagnostic Test: Antibody titration
- Covid 19 negative patients (Experimental)
  Interventions: Diagnostic Test: Blood group determination; Diagnostic Test: Antibody titration
- Untested healthy volunteers (Experimental)
  Interventions: Diagnostic Test: Blood group determination; Diagnostic Test: Antibody titration; Dietary Supplement: Probiotic

INTERVENTIONS:
Diagnostic Test: Blood group determination — Determination of the blood group (ABO/LE)
Diagnostic Test: Antibody titration — Natural anti-A and anti-B antibody levels will be determined by a gel agglutination technique on the Biorad IH-500 automaton.
Dietary Supplement: Probiotic — Administration of a probiotic to healthy volunteers to determine if it increases the level of circulating natural anti-A and anti-B antibodies (Probactiol Plus (Metagenics)).
  Arms: Untested healthy volunteers

SUMMARY:
When the COVID-19 virus infects a person, it enters the lung epithelial cells of its host and uses its genetic material to replicate.

The pulmonary epithelial cells of a part of the population, known as "secretors", are capable of expressing the antigens of the "ABO" system on their surface. This secretory status can be established by determining the antigens of the Lewis blood group system. When the virus replicates in an "secreting" individual, the antigens of the "ABO" system of the infected individual will be present on the surface of the viruses formed in his/her lungs.

It was shown in 2003 that the response of a given individual to the transmission of a virus depends on his/her blood group and on the antigens of the "ABO" system carried by the virus. A patient of group "O" would thus defend himself much better against a virus carrying antigens of blood group "A", the natural antibodies "anti-A" of the patient reducing the ability of the virus to bind to its specific receptor on pulmonary epithelial cells, to penetrate them to replicate itself. The first data collected in Wuhan (China) seems to confirm this hypothesis. A COVID-19 virus transmission model can therefore be established on the basis of blood groups.

In order to reduce the spread of the virus among nursing staff, it is possible to establish a preferential algorithm for patient management based on the "ABO" and "Lewis" blood groups of patients and "ABO" of nursing staff in health care units, if operational and human conditions allow.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 positive patients admitted within the CHU Brugmann Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Anti-A antibody concentration | baseline
  Anti-A antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-A antibody concentration | Day 4
  Anti-A antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-A antibody concentration | Week 1
  Anti-A antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-A antibody concentration | Week 2
  Anti-A antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-A antibody concentration | Week 3
  Anti-A antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-B antibody concentration | baseline
  Anti-B antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-B antibody concentration | Day 4
  Anti-B antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-B antibody concentration | Week 1
  Anti-B antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-B antibody concentration | Week 2
  Anti-B antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Anti-B antibody concentration | Week 3
  Anti-B antibody titration, as determined by gel agglutination on the Biorad IH-500 automated system.
Blood group | baseline
  Blood group (ABO/LE)

CONTACTS AND LOCATIONS:
Overall Officials: Hanane El Kenz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No